CLINICAL TRIAL: NCT06095323
Title: Comparing Level 1 Compression Sleeves With Routine Care in Preventing Breast Cancer-related Arm Lymphedema :An Open-label, Single-center, Randomized Controlled Phase II Clinical Trial
Brief Title: Comparing Level 1 Compression Sleeves With Routine Care in Preventing Breast Cancer-related Arm Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhenzhen Liu (Other Government)
Responsible Party: Sponsor-Investigator, Zhenzhen Liu, liuzhenzhen73@126.com, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-BCRL001
Record Dates: First submitted 2023-10-08; First posted 2023-10-23 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer-related Arm Lymphedema
Keywords: breast cancer-related arm lymphedema; bioimpedance spectroscopy; Limb circumference measurement
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic compression sleeves group (Experimental): The intervention group will wear compression sleeves for upper limbs with a pressure level of 1 (15-20mmHg) during the day for 12 months.
  Interventions: Device: compression sleeves for upper limbs with a pressure level of 1 (15-20mmHg)
- routine care group (No Intervention): The routine care group will proceed as an observation and receive standard lymphedema education during the clinical trial.

INTERVENTIONS:
Device: compression sleeves for upper limbs with a pressure level of 1 (15-20mmHg) — The intervention group will wear compression sleeves for upper limbs with a pressure level of 1 (15-20mmHg) during the day for 12 months.
  Arms: Prophylactic compression sleeves group

SUMMARY:
It is estimated that there are 420,000 newly diagnosed breast cancer patients in China in 2020. With surgery, radiotherapy, chemotherapy, endocrine, targeted therapy and other treatment methods going hand in hand, the outcome of breast cancer patients has been greatly improved. However, along with the comprehensive treatment of breast cancer, there will also be some corresponding complications, including breast cancer-related lymphedema （BCRL）， is one of the most common and serious complications. the incidence of BCRL in the patients with axillary dissection11% -57%, average 28%, Arm lymphedema seriously affect the quality of life of breast cancer patients, is known as the last kilometer of breast cancer patients to return to society. The related risk factors mainly include surgery, radiotherapy, body mass index, (BMI), etc.

Accordingly, a series of measures appeared to prevent the occurrence of BCRL, including surgical and non-surgical methods, The main surgical methods include lymphatic microsurgical preventing healing approach (LYMPHA), and axillary reverse mapping to retain arm lymph nodes.the LYMPHA technology requires skilled microsurgery technology, or multidisciplinary participation, which will prolong the operation time.The retention of arm lymph nodes may involve tumor safety.Non-surgical methods include elastic sleeve wearing, functional exercise, arm resistance training, manual drainage, etc. The manual drainage is time-consuming and requires therapist participation, and the evidence that resistance training can prevent edema is insufficient.The elastic cuff has been proven to effectively prevent the occurrence of BCRL, and it can prevent the accumulation of extracellular fluid caused by surgery, chemotherapy and radiation therapy, and gravity factors.

A randomized controlled study (CTRI / 2017 / 12 / 010762) released by Paramanandam VS et al, Tata Memorial Hospital, tertiary Cancer Center, Mumbai, India, that wearing compression sleeves (20-25mmHg) can reduce and delay the occurrence of arm swelling in the first year after breast cancer surgery. However, the higher pressure sleeves still has a negative impact on patients' quality of life and patient compliance. Ochalek K have shown that the primary pressure sleeves (15-20mmHg) is also effective in preventing the occurrence of lymphedema, but the randomized controlled study has a small sample size and insufficient evidence.

DETAILED DESCRIPTION:
It is estimated that there are 420,000 newly diagnosed breast cancer patients in China in 2020. With surgery, radiotherapy, chemotherapy, endocrine, targeted therapy and other treatment methods going hand in hand, the outcome of breast cancer patients has been greatly improved. However, along with the comprehensive treatment of breast cancer, there will also be some corresponding complications, including breast cancer-related lymphedema （BCRL）， is one of the most common and serious complications. the incidence of BCRL in the patients with axillary dissection11% -57%, average 28%, Arm lymphedema seriously affect the quality of life of breast cancer patients, is known as the last kilometer of breast cancer patients to return to society. The related risk factors mainly include surgery, radiotherapy, body mass index, (BMI), etc.

Accordingly, a series of measures appeared to prevent the occurrence of BCRL, including surgical and non-surgical methods, The main surgical methods include lymphatic microsurgical preventing healing approach (LYMPHA), and axillary reverse mapping to retain arm lymph nodes.the LYMPHA technology requires skilled microsurgery technology, or multidisciplinary participation, which will prolong the operation time.The retention of arm lymph nodes may involve tumor safety.Non-surgical methods include elastic sleeve wearing, functional exercise, arm resistance training, manual drainage, etc. The manual drainage is time-consuming and requires therapist participation, and the evidence that resistance training can prevent edema is insufficient.The elastic cuff has been proven to effectively prevent the occurrence of BCRL, and it can prevent the accumulation of extracellular fluid caused by surgery, chemotherapy and radiation therapy, and gravity factors.

A randomized controlled study (CTRI / 2017 / 12 / 010762) released by Paramanandam VS et al, Tata Memorial Hospital, tertiary Cancer Center, Mumbai, India, that wearing compression sleeves (20-25mmHg) can reduce and delay the occurrence of arm swelling in the first year after breast cancer surgery. However, the higher pressure sleeves still has a negative impact on patients' quality of life and patient compliance. Ochalek K have shown that the primary pressure sleeves (15-20mmHg) is also effective in preventing the occurrence of lymphedema, but the randomized controlled study has a small sample size and insufficient evidence. This study aims to compare level 1 compression sleeves with routine care in preventing breast cancer-related arm lymphedema after axillary lymph node dissection through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years old
2. Breast cancer, unilateral，Patients undergoing axillary lymph node dissection
3. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. arm swelling preoperatively, as assessed by bioimpedance spectroscopy (BIS) or Limb circumference measurement
2. any condition that hindered them from wearing a compression sleeve
3. Patients with upper limb dysfunction before surgery, including shoulder and elbow joint mobility disorders
4. Patients with mental disorders, senile dementia, and cognitive impairments，were not able to complete a questionnaire independently
5. Patients with bilateral breast cancer, recurrence, or metastasis to other organs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of arm lymphedema 2 years after surgery: as assessed by bioimpedance spectroscopy (BIS) | Preoperatively ，postoperatively 3、6、9、12、18、24 month
  Incidence of arm lymphedema 2 years after surgery: as assessed by bioimpedance spectroscopy (BIS), bilateral upper limb impedance ratio, bilateral upper limb impedance ratio compared with the first baseline, if the inter-arm ratio exceeds the threshold, the individual is classified as arm lymphedema . If the surgical side is the dominant hand, the inter-arm impedance ratio threshold is 1.108; if the non-dominant hand is used, the inter-arm impedance ratio threshold is 1.072.

SECONDARY OUTCOMES:
Incidence of arm lymphedema 2 years after surgery: as assessed by circumferential diameter measureme | Preoperatively ，postoperatively 3、6、9、12、18、24 month
  Arm vol-ume was determined from circumference measurements,commencing at the ulnar styloid and at 10-cm intervals proximally to 40 cm using an inelastic tape measure; measurements were recorded to the nearest 1.0 mm. Each arm's volume was calculated using the truncated cone formula from the arm circumference measurements.Relative (percentage) arm volume differences between the at-risk and unaffected arms were then calculated, and cases in which the relative arm volume increased 10% from baseline were identified.
the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the breast cancer-specific (BR23) questionnaire | Preoperatively ，postoperatively 3、6、9、12、18、24 month
  the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and the breast cancer-specific (BR23) questionnaire was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No